CLINICAL TRIAL: NCT05941832
Title: ASM in CF:ANNE Sensor Monitoring in Cystic Fibrosis
Brief Title: ANNE Sensor Monitoring in Cystic Fibrosis
Acronym: ASM in CF
Status: Completed | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: LifeArc (Other); Cystic Fibrosis Trust (Other)
Responsible Party: Sponsor
Other Study IDs: P02784
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: ANNE Chest Sensor — Wearing ANNE Chest Sensor for 6 weeks

SUMMARY:
The ANNE sensor is a small, wire free device that is placed on the chest with a removable adhesive patch. It measures things like temperature, heart rate and breathing rate without the need for wires and large machines that are needed currently. The aim is to trial this sensor in a small group of participants to see how well it is tolerated and how well it measures. The aim is to see if the sensor could provide additional information to help the medical team detect when a participant is becoming unwell with less need for the participant to perform repeated tests.

Participants will wear the sensor for 6 weeks continuously (apart from when it is charged for 4-6 hours each day). Participants can perform their usual activities whilst wearing the sensor but should not submerse the sensor in water for long periods of time.

DETAILED DESCRIPTION:
Rationale

The aim of this study is to explore the potential use of the ANNE Chest Sensor to assist or improve the detection of health conditions in people with CF. The emphasis is on identifying onset and progression of pulmonary exacerbations.

The ANNE Chest Sensor is now being applied to help people with respiratory and other conditions. Through advanced analytics and signal processing, the device includes an accelerometer, temperature sensor and electrocardiogram, from which vital signs such as respiratory rate, skin and body temperature, ECG, heart rate, step count, fall count and body position can be measured.

Royal Papworth Hospital has demonstrated that daily recordings of a range of physiological parameters (e.g., spirometry, pulse oximetry, activity, heart rate, etc.) in combination with self-reported survey responses (e.g., general wellness, cough, sleep quality) in people with CF holds promise to more accurately track fluctuations in health condition(s), in particular the start of pulmonary exacerbations (PE). This data is collected remotely at the study participant's home using remote/virtual online tools, as part of a larger effort to take a more virtual approach to clinics. Passive and continuous collection of a patient's data for early detection is a natural extension of this approach.

Study Design

This is a 6-month single-centre observational, prospective study, designed as a pilot study. We aim to recruit 10 adult patients with Cystic Fibrosis (CF) who are already participating in the Project Breathe home monitoring project at Royal Papworth Hospital. Participants will be enrolled for 6 weeks.

This study is designed to run as a non-disruptive study with no impact on routine clinical care and the sensor data will have no influence on treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cystic Fibrosis based on genetic testing and /or sweat chloride levels.
* At least >/= 18 years of age at time of consent
* Able to provide written informed consent
* Patients who are currently undertaking home monitoring / virtual clinics as part of Project Breathe

Exclusion Criteria:

* Patients unable to provide written informed consent
* Patients who are currently not undertaking home monitoring / virtual clinics as part of Project Breathe
* Lung transplant recipients.
* Severe skin conditions e.g. psoriasis, severe eczema
* Patients with a pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Cystic Fibrosis who are being treated at Royal Papworth Hospital Cystic Fibrosis Specialist Centre.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With ANNE Sensor Related Adverse Skin Sensitivity Events | 6 weeks
  Number of ANNE sensor related Adverse Events reported during the study

SECONDARY OUTCOMES:
Difference in Heart Rate (bpm) Measured by The ANNE Chest Sensor vs Current Heart Rate Home Monitoring | 6 weeks
  Number of beats per minute (bpm) measured by the ANNE Chest Sensor vs current home heart rate monitoring (bpm)
Difference in Oxygen Levels (%) Measured by The Anne Chest Sensor vs Current Oxygen Levels Home Measurements | 6 weeks
  Blood oxygen levels (%) measured by the ANNE Chest Sensor vs current home oxygen level monitoring (%)
Difference in Activity (kcal) Measured by The ANNE Chest Sensor vs Current Home Activity Monitoring | 6 weeks
  Kcal expended through exercise as measured by the ANNE Chest Sensor vs current home monitoring of activity (kcal)

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Papworth Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This is undecided currently